CLINICAL TRIAL: NCT00766441
Title: Sitagliptin Versus Sulphonylurea Based Treatments in Muslim Patients With Type 2 Diabetes During Ramadan
Brief Title: Sitagliptin Versus Sulphonylurea in Type 2 Diabetes During Ramadan
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: inadequate recruitment
Sponsor: University of Manchester (Other)
Responsible Party: Professor R A Malik, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08/H1005/46
Record Dates: First submitted 2008-10-03; First posted 2008-10-06 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2008-10

CONDITIONS: Diabetes; Hypoglycemia
Keywords: diabetes; hypoglycemia; ramadan; fasting
MeSH Terms: conditions — Diabetes Mellitus; Hypoglycemia; Fasting | interventions — Sitagliptin Phosphate; Sulfonylurea Compounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Sitagliptin 100mg
  Interventions: Drug: Sitagliptin
- 2 (Active Comparator): Sulphonylurea
  Interventions: Drug: sulphonylurea

INTERVENTIONS:
Drug: Sitagliptin — tablet, 100mg, once daily, 4 weeks
  Arms: 1
Drug: sulphonylurea — sulphonylurea, variable, od or bd, during ramadan
  Arms: 2

SUMMARY:
This study will assess if Sitagliptin addition to metformin or glitazone is better than current sulphonylurea based treatments during Ramadan. The rationale is that Sitagliptin offers metabolic advantages primarily with the low incidence of hypoglycemia over current sulphonylurea based treatments.

DETAILED DESCRIPTION:
To define metabolic alterations during Ramadan:

1. Primary end point: Occurrence of hypoglycemia. The patients will record hypoglycaemic episodes in a self-monitoring diary together with blood glucose values.
2. Secondary endpoints: Body weight, fasting blood sugar (FBS), glycosylated haemoglobin (HbA1c)/Fructosamine, triglycerides (TG), total cholesterol (TC), low-density lipoprotein-cholesterol (LDL-C) and high density lipoprotein-cholesterol (HDL-C).
3. A subgroup will undergo CGMS assessment to define glycaemic excursions during and after fasting.

ELIGIBILITY:
Inclusion Criteria:

1. Muslim men and women with Type 2 diabetes.
2. Age 18-78 years
3. Intending to fast during the month of Ramadan
4. On oral antihyperglycemic agents (sulphonylurea based/combination therapy)

Exclusion Criteria:

1. Patient with hypersensitivity or contraindication to Sitagliptin treatment
2. Patient with CKD (creatinine clearance <50 ml/min)
3. Patients who have participated in another intervention study in the last 2 months
4. Patients who do not give informed consent
5. Pregnant or breast feeding women.
6. Patients on insulin
7. Patients with severe liver disease

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-08; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Occurrence of hypoglycemia | 4 weeks during Ramadan

SECONDARY OUTCOMES:
Body weight, fasting blood sugar, HbA1c, triglycerides, total cholesterol, LDL-C, HDL-C. CGMS to define glycaemic excursions | 4 weeks during Ramadan

CONTACTS AND LOCATIONS:
Overall Officials: Rayaz A Malik, MBChB, PhD, Principal Investigator — University of Manchester
Locations (1):
- Wellcome Trust Clinical Research Facility, Manchester, United Kingdom